CLINICAL TRIAL: NCT00000594
Title: NHLBI Type II Coronary Intervention Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 400
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Hypercholesterolemia, Familial; Myocardial Infarction; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Hyperlipoproteinemia Type II; Myocardial Infarction; Myocardial Ischemia | interventions — Cholestyramine Resin

INTERVENTIONS:
Drug: cholestyramine

SUMMARY:
To determine whether lowering of cholesterol with cholestyramine in a population with Type II hyperlipidemia led to a decreased rate of progression (a regression of coronary artery disease) as demonstrated by death, myocardial infarction, or progression of disease on angiography.

DETAILED DESCRIPTION:
BACKGROUND:

There is overwhelming evidence that increased cholesterol levels are associated with increased risk of cardiovascular disease. This study examined whether lowering of cholesterol through drug therapy in people who had coronary artery disease as determined by angiography led to regression of the disease, again as indicated by angiography and reduction in mortality or nonfatal myocardial infarction. The study should be contrasted with the Coronary Primary Prevention Trial (CPPT), which determined whether lowering cholesterol through a combination of drug and diet therapy resulted in decreased cardiovascular mortality. It should be noted that patients in the CPPT did not have known preexisting coronary heart disease.

DESIGN NARRATIVE:

A randomized, double-blind trial, with single experimental and control groups. The experimental group received drug therapy (cholestyramine); the control group received placebo. Both groups received diet therapy. The endpoints were a significant difference in the progression of coronary disease as shown by angiography or a significant difference in new myocardial infarction or death. Patients were followed under therapy for at least 5 years.

ELIGIBILITY:
Men and women with angiographically demonstrated coronary artery disease.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1971-11; Study Completion 1976-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Brensike — Cardiology Branch, NHLBI

REFERENCES:
- [Background] Borer JS, Brensike JF, Redwood DR, Itscoitz SB, Passamani ER, Stone NJ, Richardson JM, Levy RI, Epstein SE. Limitations of the electrocardiographic response to exercise in predicting coronary-artery disease. N Engl J Med. 1975 Aug 21;293(8):367-71. doi: 10.1056/NEJM197508212930801. PMID 168493
- [Background] Belmaker RH, Pollin W, Jenkins CD, Brensike J. Coronary prone behavior pattern in a sample of type II hypercholesteremic patients. J Psychosom Res. 1976;20(6):591-4. doi: 10.1016/0022-3999(76)90061-1. No abstract available. PMID 190398
- [Background] Aldrich RF, Brensike JF, Battaglini JW, Richardson JM, Loh IK, Stone NJ, Passamani ER, Ackerstein H, Seningen R, Borer JS, Levy RI, Epstein SE. Coronary calcifications in the detection of coronary artery disease and comparison with electrocardiographic exercise testing. Results from the National Heart, Lung, and Blood Institute's type II coronary intervention study. Circulation. 1979 Jun;59(6):1113-24. doi: 10.1161/01.cir.59.6.1113. No abstract available. PMID 582024
- [Background] Brensike JF, Kelsey SF, Passamani ER, Fisher MR, Richardson JM, Loh IK, Stone NJ, Aldrich RF, Battaglini JW, Moriarty DJ, Myrianthopoulos MB, Detre KM, Epstein SE, Levy RI. National Heart, Lung, and Blood Institute type II Coronary Intervention Study: design, methods, and baseline characteristics. Control Clin Trials. 1982 Jun;3(2):91-111. doi: 10.1016/0197-2456(82)90038-1. PMID 6749427
- [Background] Brensike JF, Levy RI, Kelsey SF, Passamani ER, Richardson JM, Loh IK, Stone NJ, Aldrich RF, Battaglini JW, Moriarty DJ, et al. Effects of therapy with cholestyramine on progression of coronary arteriosclerosis: results of the NHLBI Type II Coronary Intervention Study. Circulation. 1984 Feb;69(2):313-24. doi: 10.1161/01.cir.69.2.313. PMID 6360414
- [Background] Levy RI, Brensike JF, Epstein SE, Kelsey SF, Passamani ER, Richardson JM, Loh IK, Stone NJ, Aldrich RF, Battaglini JW, et al. The influence of changes in lipid values induced by cholestyramine and diet on progression of coronary artery disease: results of NHLBI Type II Coronary Intervention Study. Circulation. 1984 Feb;69(2):325-37. doi: 10.1161/01.cir.69.2.325. PMID 6360415
- [Background] Brown BG, Lin JT, Kelsey S, Passamani ER, Levy RI, Dodge HT, Detre KM. Progression of coronary atherosclerosis in patients with probable familial hypercholesterolemia. Quantitative arteriographic assessment of patients in NHLBI type II study. Arteriosclerosis. 1989 Jan-Feb;9(1 Suppl):I81-90. PMID 2912435